CLINICAL TRIAL: NCT03616054
Title: INternational Observational Study To Understand the Impact and BEst Practices of Airway Management in Critically Ill Patients
Brief Title: International Observational Study on Airway Management in Critically Ill Patients
Acronym: INTUBE
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera San Gerardo di Monza (Other)
Responsible Party: Principal Investigator, Vincenzo Russotto, MD, MD, Azienda Ospedaliera San Gerardo di Monza
Other Study IDs: INTUBE
Record Dates: First submitted 2018-07-15; First posted 2018-08-06 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Critical Illness; Respiratory Failure; Hemodynamic Instability; Coma
Keywords: Airway management
MeSH Terms: conditions — Critical Illness; Respiratory Insufficiency; Coma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endotracheal intubation (ETI) is a potentially life-threatening procedure for critically ill patients and major severe complications such as severe hypoxia, cardiovascular collapse and cardiac arrest are common. Despite the high risk of the procedure, different interventions lack high-quality evidence and the investigators hypothesize that a heterogeneous practice among different centres and geographical areas may be found.

The investigators designed a large international observational study aiming at prospectively collecting data on the current impact of ETI-related adverse events and current airway management practice in critically ill patients. Investigators will collect data on all consecutive in-hospital (intensive care unit, emergency department and wards) ETIs performed in adult critically patients.

DETAILED DESCRIPTION:
This study aims at prospectively collecting data on the current morbidity and mortality of ETI-related adverse events and current airway management practice in adult critically ill patients. Investigators designed a large international study calling for participation all institutions caring critically ill patients worldwide.

Inclusion criteria

Investigators will include all adult (≥ 18 years old) critically ill patients undergoing intubation during the period of observation. Investigators will consider all in-hospital intubations. Critically ill will be defined those patients with a life-threatening condition requiring intubation for either cardiorespiratory failure or airway protection.

Exclusion Criteria

* Intubation performed in the out-of-hospital setting
* Intubation during cardiac arrest
* Intubation performed for anaesthesia

Primary Outcome

Major ETI-related adverse events - composite outcome (severe hypoxemia, cardiac arrest and cardiovascular collapse - see further for definitions)

Secondary Outcomes

Minor ETI-related adverse events and ICU mortality (see further for definitions).

Sample size

Investigators' aim is to collect data from 1000 intubation- related major complications. From a previously published report (Jaber 2006) the expected incidence of at least one major complication is 28%. Therefore investigators plan to recruit data from 3600 endotracheal intubations. Intubation rate may vary from 0.5 to 2 ETIs/day according to different centres (e.g. total hospital beds, number of ICUs and ICU beds) and local policies. Each centre will be asked to collect data from 20 ETIs. A maximum time window of 8 weeks will be allowed for each centre (i.e. for centres with a slower recruitment rate, data collection will stop after 8 weeks irrespective of total number of ETIs collected data). Investigators plan to recruit at least 180 centres worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients undergoing in-hospital endotracheal intubation.

Exclusion Criteria:

* Intubation performed in the out-of-hospital setting;
* Intubation during cardiac arrest;
* Intubation performed only for anaesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will include all adult (≥ 18 years old) critically ill patients undergoing intubation during the period of observation. We will consider all in-hospital intubations. We will define critically ill those patients with a life-threatening condition requiring intubation for either cardiorespiratory failure or airway protection.
Sampling Method: Probability Sample
Enrollment: 3600 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Major intubation-related complication | 30 minutes
  At least one of the following (composite outcome):
  * Severe hypoxemia (SpO2 < 80%) occurring within 30 minutes from intubation
  * Cardiac arrest occurring within 30 minutes from intubation
  * Cardiovascular collapse (at least one of the following), occurring within 30 minutes from intubation:
    * Systolic arterial pressure < 65 mmHg recorded 1 time
    * SAP < 90 mmHg for > 30 minutes
    * New need of vasopressors/their increase and/or fluid load > 15 ml/kg to maintain the target blood pressure.

SECONDARY OUTCOMES:
Cardiac arrhythmia | 30 minutes
  New onset of any supraventricular or ventricular arrhythmia
Difficult intubation | 30 minutes
  > 2 laryngoscopic attempts
Cannot intubate cannot oxygenate scenario (CICO) | 30 minutes
  'Oxygenation' cannot be achieved using the anatomical conduits of the upper airway
Emergency front of neck airway (FONA) | 30 minutes
  Cricothyroidotomy, percutaneous tracheostomy, surgical tracheostomy
Aspiration of gastric contents | 24 hours
  Inhalation of oro-pharyngeal or gastric contents into the larynx and the respiratory tract
Oesophageal intubation | 30 minutes
  Accidental placement of endotracheal tube into the oesophagus
Pneumothorax/pneumo-mediastinum | 24 hours
  Pleural/mediastinal air collection attributable to traumatic airway management
Dental injury | 24 hours
  Any notable change to the patient's dentition attributable to the procedure of endotracheal intubation
Airways injury | 24 hours
  Any detectable/clinically relevant airways injury attributable to the endotracheal intubation procedure (e.g.bleeding, tracheal tear/laceration)
ICU mortality | up to 12 weeks
  Survival status at ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Russotto, MD, Principal Investigator — Department of Emergency and Intensive Care, University Hospital San Gerardo Monza, ASST Monza, Monza, Italy; Giacomo Bellani, MD, PhD, Principal Investigator — Department of Emergency and Intensive Care, University Hospital San Gerardo Monza, ASST Monza, Monza, Italy; University of Milano Bicocca
Locations (1):
- ASST Monza - University Hospital San Gerardo, Monza, Italy

REFERENCES:
- [Derived] Russotto V, Laffey JG, Tassistro E, Myatra SN, Rezoagli E, Foti G, Antolini L, Valsecchi MG, Bauer PR, Szuldrzynski K, Camporota L, Greif R, Higgs A, Parotto M, Fumagalli R, Sorbello M, Robba C, Grasselli G, Bellani G, Caironi P, Lascarrou JB; INTUBE Study Investigators. Peri-intubation complications in critically ill obese patients: a secondary analysis of the international INTUBE cohort. Crit Care. 2025 May 13;29(1):192. doi: 10.1186/s13054-025-05419-2. PMID 40361245
- [Derived] Russotto V, Lascarrou JB, Tassistro E, Parotto M, Antolini L, Bauer P, Szuldrzynski K, Camporota L, Putensen C, Pelosi P, Sorbello M, Higgs A, Greif R, Grasselli G, Valsecchi MG, Fumagalli R, Foti G, Caironi P, Bellani G, Laffey JG, Myatra SN; INTUBE Study Investigators. Efficacy and adverse events profile of videolaryngoscopy in critically ill patients: subanalysis of the INTUBE study. Br J Anaesth. 2023 Sep;131(3):607-616. doi: 10.1016/j.bja.2023.04.022. Epub 2023 May 17. PMID 37208282
- [Derived] Russotto V, Tassistro E, Myatra SN, Parotto M, Antolini L, Bauer P, Lascarrou JB, Szuldrzynski K, Camporota L, Putensen C, Pelosi P, Sorbello M, Higgs A, Greif R, Pesenti A, Valsecchi MG, Fumagalli R, Foti G, Bellani G, Laffey JG. Peri-intubation Cardiovascular Collapse in Patients Who Are Critically Ill: Insights from the INTUBE Study. Am J Respir Crit Care Med. 2022 Aug 15;206(4):449-458. doi: 10.1164/rccm.202111-2575OC. PMID 35536310